CLINICAL TRIAL: NCT05960747
Title: Improvement to Perform Thoracocentesis After a Specific Training in Medical Students With the Supervised Use of an Augmented Reality Simulator
Acronym: ARPEGES
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8809
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pleural Effusion; Frist Time Indication to Perform a Thoracentesis; Medical Student Training
Keywords: Thoracentesis; Augmented virtual reality simulator; Medical student training
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: Medical students with standard training: theoretical teaching, associated with a real-life demonstration of at least one thoracentesis by a senior doctor from our department
- Simulation group: Medical students with standard training + training using an augmented virtual reality simulator specially developed for thoracentesis.
  Interventions: Other: Simulation group

INTERVENTIONS:
Other: Simulation group — Specific training for medical students by using an augmented virtual reality simulator for thoracentesis
  Groups: Simulation group

SUMMARY:
Monocentric study, aiming to assess the improvement of medical students to perform a first-time thoracentesis after training using a specific training using an augmented virtual reality simulator, versus standard training.

Study population: medical students from the department of Respirology (University hospital of Strasbourg), performing their first thoracocentesis in patients having an indication for a first-time thoracocentesis.

This is not an interventional study, no change in patient course being induced because of the study.

After the procedure: use of specific surveys for the patient and for medical students to assess the patient's pain, the patient and the medical student level of anxiety, and the student ability during the procedure.

ELIGIBILITY:
Medical students :

Inclusion criteria:

* Medical students between the 4th and 6th year of their medical course, working in the department of respirology at the University hospital of Strasbourg, France, without any prior experience of thoracocentesis.
* Older than 18 years old
* No opposition to participate to the study (signed consent form).

Exclusion criteria:

- Student with a prior experience of pleural procedure (chest tube, thoracocentesis).

Patients :

Inclusion criteria:

* Patients requiring a first-time thoracentesis in routine care.
* Older than 18 years old.
* Speaking and understanding French.
* Valid health insurance.
* No opposition to participate to the study (signed consent form).

Exclusion criteria:

* Patient with previous experience of pleural procedure (thoracocentesis, chest tube…).
* Patient having a high-volume pleural effusion according to radiological/ultrasound criteria.
* Patient with low-volume pleural effusion according to radiological/ultrasound criteria.
* Patient with poor clinical tolerance of the pleural effusion(respiratory instability, dependence on ventilation machine with positive expiratory pressure…).
* Patients with higher risk of complication during the procedure (BMI > 35 kg/m², with increased risk of bleeding…).
* Contraindication to the use of Lidocaine.
* Local infection.
* Impossibility to provide detailed information to the patient.
* Subject under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Medical students between the 4th and 6th year of their medical course, working in the department of respirology at the University hospital of Strasbourg, France, without any prior experience of thoracocentesis.
  * Patients requiring a first-time thoracentesis in routine care
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of the success rate | 1 day
  Assessment of the success rate to perform a first-time thoracentesis in patients with an indication for this procedure, depending on whether the medical student was trained using an augmented virtual reality simulator, or with standard training

SECONDARY OUTCOMES:
Assessment of specific characteristic prior and after thoracocentesis | 1 day
  Assessment of specific characteristic prior and after thoracocentesis for the patient (pain, anxiety), and for the medical student (theorical knowledge, anxiety, ability during the procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopitaux Universitaire de Strasbourg, Strasbourg, Bas-Rhin
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided